CLINICAL TRIAL: NCT06148896
Title: Effects of Combining Physiotherapy Group Exercise With Acceptance and Commitment Therapy in Elderly With Chronic Nonspecific Low Back Pain: A Randomized Controlled Trial
Brief Title: Combining Physiotherapy Group Exercise With Acceptance and Commitment Therapy in Elderly With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT_YKC
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-11

CONDITIONS: Chronic Low Back Pain
Keywords: Elderly; Chronic non specific low back pain; Group exercise; Acceptance and Commitment therapy led by physiotherapist

STUDY DESIGN:
Intervention Model Description: This two-armed randomised controlled trial (RCT) aims to investigate the effectiveness of Group Exercise with PACT (GrExPACT experimental intervention) as compared to Group Exercise (GrEx) alone led by physiotherapist (control intervention) for elderly with chronic LBP
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be blinded by informing them that they will participate in one of the two treatment groups that is known to be helpful to their chronic nonspecific back pain but not known which one is better. An independent assessor who is responsible for carrying out the physical test and assist the elderly in filling of the questionnaires will be blinded for the group allocation. The research personnel who is responsible for data entry and statistical analysis will also be blinded for the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Exercise with acceptance and commitment therapy (Experimental): Combining physiotherapy group exercise with acceptance and commitment therapy delivered by physiotherapist (GrExPACT)
  Interventions: Behavioral: GrExPACT
- Group Physiotherapy Exercise alone (Active Comparator): Group Physiotherapy exercise alone (GrEx)
  Interventions: Behavioral: GrEx

INTERVENTIONS:
Behavioral: GrExPACT — Combining physiotherapy group exercise with acceptance and commitment therapy delivered by physiotherapy
  Other Names: No other intervention (No drug, No device)
  Arms: Group Exercise with acceptance and commitment therapy
Behavioral: GrEx — Group physiotherapy exercise
  Other Names: No other intervention (No drug, No device)
  Arms: Group Physiotherapy Exercise alone

SUMMARY:
This two-armed randomized controlled trial (RCT) aims to investigate the effectiveness of Group Exercise with acceptance and commitment therapy led by physiotherapist (GrExPACT) (experimental intervention) as compared to Group Exercise alone (GrEx) (control intervention) for elderly with chronic low back pain (LBP) whom are stratified as medium or high-risk using the STarT Back Screening Tool on functional recovery as measured by Roland Morris Disability Questionnaire as the primary outcome and a list of secondary outcomes which include Committed Action questionnaire, Chronic Pain Acceptance questionnaire, Patient self-efficacy Questionnaire, Brief Pain Inventory, Patient Specific Functional Scale, Short Physical Performance Battery and a patient satisfaction survey, immediately after a 5-week programme as well as at 3-month follow-up.

The list of hypotheses to be tested in this RCT include:

1. For main effect: Intervention H0: The outcome means for the intervention of GrExPACT and GrEx are equal H1: The outcome means for the intervention of GrExPACT and GrEx are not equal
2. For main effect: Time H0: The outcome means for the time with measuring point at pre-intervention, immediate after the program and at 3 months are equal H1: The outcome means for the time with measuring point at pre-intervention, immediate after the program and at 3 months are not equal
3. For interaction: Intervention x Time H0: There is no interaction between the intervention and time H1: There is interaction between the intervention and time

DETAILED DESCRIPTION:
Sample size:

The sample size was calculated with reference to the effect size of 0.052 (partial eta square) being worked out from the primary outcome of Roland Morris Disability Questionnaire obtained from the pilot study. G*Power 3.1.9.4 was used to calculate the sample size. With power of 0.95 and alpha value of 0.05, the total sample size is 68. With reference to the attrition rate of approximately 20% in the pilot study, the sample size will become 43 subjects in each group and with total of 86 subjects will be recruited.Subjects will be recruited from local community elderly community centers.

Randomization:

The subjects will be randomly assigned by the principal investigator to either intervention group of GrExPACT or control group of GrEx using computerized randomization software. Permuted blocked randomization with a block size of four and stratified by gender and STarT Back category will be used as to ensure the groups are balanced. The allocation will be concealed and stored in an encrypted file storing in a password protected computer. Corresponding group therapy class will be arranged to the patient accordingly.

Study design:

86 subjects with chronic nonspecific LBP subject will first receive a 30-minute triage screening by a physiotherapist for inclusion criteria, exclusion criteria and red flags as to confirm the subjects are belonging to chronic nonspecific LBP and is suitable for the study. The red flags include night pain, 24-hour pain, unexplained weight loss, night sweats, fever, change in bowel and urinary habits and saddle anesthesia. Subjective examination for body chart and physical examination include trunk range of motion, myotome, dermatome, reflexes, palpation, and neuro-tension test will be performed when applicable.

Each subject will participate weekly group program for five consecutive weeks after the group randomization. The size of the group is about 10. Each session for both intervention group and control group will last for 105 min and will receive 60-minute group exercise therapy includes supervised stretching, mobilization, stabilization and strengthening exercise for the muscles around lumbar, hips and low limbs followed by functional and aerobic training. The exercises are selected with reference to the National Institute for health and care Excellence (NICE) guidelines, systematic review for physical activities for elderly with chronic LBP and experience from the previous pilot trial which is safe and effective for elderly with nonspecific chronic LBP. The exercise will be taught to patient progressively from lying to sitting in first two sessions and adding more advance standing to functional and aerobic training in subsequent sessions. The resistance of the TheraBand and step height for functional training will tailor made and increase according to individual capability. Each patient will be given an exercise pamphlet, goal setting worksheet and home exercise record sheet. Patients are encouraged to utilize local community exercise facilitates and bring back the home exercise record sheet each time for checking of compliance of practicing home exercise.

Both groups of patients will have a physiotherapist leading discussion. For the GrEx group, the discussion will last for 45 minutes. It involves discussion for back care and exercise referencing to the back school that is a common educational and training program given to patients with low back pain. The content includes anatomy of the spine, cause for pain, self-management, correct manual lifting technique, ergonomic advice, and benefit of regular exercise. For the GrExPACT group, the discussion will use the Acceptance and Commitment Therapy (ACT) approach and will also last for 45 minutes. The content of the discussion will follow the protocol-based ACT extracted from the protocol for the contextual pain management by physiotherapy being used in INPUT center of St Thomas Hospital, London and physiotherapy informed by acceptance and commitment therapy protocol (PACT) .

Qualification of the intervention provider:

The intervention providers are registered physiotherapist in Hong Kong who had more than 30 years of clinical experience in treating patient with musculoskeletal problem at public physiotherapist outpatient clinic. For the background of ACT training, the physiotherapists had received training for taught course for ACT and had participated in a two-day clinical attachment for the contextual pain management program in INPUT Center at St. Thomas Hospital in London of United Kingdom in 2018. Besides the participation in the local pilot trial for GrExPACT study, they had also participated in the development for the local clinical service team for stratified care and combined the physical and psychological approach in management of high-risk back pain patients since 2015.

Data processing and statistical analysis:

The statistical analysis will be carried out using IBM SPSS version 28 software. The demographically data will be presented by descriptive statistics. For continuous data, it will be presented as mean, standard deviation and range. For categorical data, it will be presented as frequency and percentage. Normality will be first screened by Boxplot, and further assessed by the Shapiro-Wilk test. For the primary and secondary outcomes, two way repeated measure ANOVA will be carried out. For the effect of time, the post hoc test will be carried out for testing the differences of outcome scores for pre-intervention verse immediate after the program; pre-intervention verse at 3 months; and immediate after the program verse at 3 months. For the effect of intervention, post hoc tests at each time point will be carried out when necessary. Significance was set at p < 0.05. Intention-to-treat analysis will be used and missing data will be replaced with data from the nearest previous non-missing data. Effect sizes (Partial eta squared) will also be computed to establish the magnitude of the treatment effects. The effect sizes will interpreted as small (η2=0.01), medium (η2=0.06) or large (η2=0.14).

Clinical significance:

In the management of elderly patient with chronic nonspecific low back pain (LBP), to face the aging population, growing high patient volume and limited resources in health care, an effective and efficient service model is urged. The service model of GrExPACT in the present randomized control trial involve tailor made and resources saving strategy by using concept of stratified care with STarT Back Screening Tool, physical therapy with group exercise and psychological therapy with group ACT lead by physiotherapist. With the present study, the effectiveness, synergistic effect, and adaptability to local culture for combining physiotherapy group exercise with acceptance and commitment therapy delivered by physiotherapist (GrExPACT) could be studied. The potential positive finding may enhance the role of physiotherapist using the psychological approach in the management of chronic nonspecific LBP and provide evidence support for the proposed more comprehensive, tailor made and resources saving service model of GrExPACT. This may help to reform a more effective and efficient model of care in Hong Kong.

ELIGIBILITY:
Inclusion Criteria

1. Ages ≥ 65;
2. Nonspecific LBP for > 3 month;
3. Stratified as medium-risk category (i.e., total score ≥ 4 and sub score ≤ to 3) and high-risk category (i.e., total score ≥ 4 and sub score ≥ 4) using the STarT Back Screening Tool;
4. Roland Morris Disability Questionnaire (RMDQ) score ≥ 5 (with reference to the minimal level of detectable change)(30, 31);
5. Able to walk with or without assistive aid and with Modified Functional Ambulatory Category ≥ 6 (32);
6. Able to read Chinese characters;
7. Able to speak and understand Cantonese; and
8. Abbreviated mental test (AMT) ≥ 6 (33).

Exclusion Criteria

1. Specific cause of LBP such as tumor, infection, or apparent neurological deficit;
2. Serious uncontrolled co-morbidities or systematic diseases which is contraindicated to exercise;
3. Orthopedic condition like recent fracture require immobilization and not fitting for exercise;
4. Unstable cardiac, pulmonary, metabolic, and psychological disease requiring acute care;
5. Severe cognitive, language or hearing deficits;
6. Spinal surgery in the past 12 months as not to confound with effect of surgery;
7. People who had prior treatment with ACT at any time; or
8. People who had received physiotherapy treatment in the previous 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire | Pre-intervention, immediate post-intervention and 3 month post-intervention
  The Roland Morris Disability Questionnaire is a 24 self-administrated items scale which measures the level of disability of patients with LBP. Items are yes and no response in which the item will score 0 with negative response and score 1 for positive response. The score for the Roland Morris Disability Questionaire is the sum of scores of the items with positive response. A patient score can range from 0 to 24. The higher the score, the greater is the disability.

SECONDARY OUTCOMES:
Committed Action Questionnaire | Pre-intervention, immediate post-intervention and 3 month post-intervention
  The Committed Action Questionnaire is a self-reported 8 item questionnaire assessing the construct of committed action from the psychological flexibility model of Acceptance and Commitment Therapy. It composed of two subscales naming values persistence which consist of 4 positively keyed items and nonreactive behavior which consist of 4 negatively keyed items. Each items requires to rate with a 7-point Likert scale ranging from 0 (never true) to 6 (always true). The score for items being negatively keyed need to be reversed before calculation of the total score. The sum of score for the eight items forming a total score ranging from 0 to 48. The higher the total scores the greater the committed action.
Chronic Pain Acceptance Questionnaire | Pre-intervention, immediate post-intervention and 3 month post-intervention
  The Chronic Pain Acceptance Questionnaire 8 is a self-reported 8-item questionnaire used to measure the acceptance of pain. It composed of two subscales naming activity engagement and pain willingness. The 4 item under activity engagement evaluates the degree to which behaviors are limited or restricted by pain. The 4 item under pain willingness assesses the degree of effort directed at controlling pain. Each items requires to rate with a 7-point Likert scale ranging from 0 (never true) to 6 (always true). The score for the items under the subscale of pain willingness need to be reversed before calculation of the score. The sum of score for the eight items forming a total score ranging from 0 to 48. The higher the total scores the greater levels of pain acceptance.
Pain self-efficacy Questionnaire | Pre-intervention, immediate post-intervention and 3 month post-intervention
  Pain self-efficacy Questionnaire (PSEQ) is a self-reported 10-item questionnaire to evaluate the confidence of people with chronic pain to perform activities such as household chores, work and social activities while in pain. Each item needs to rate with a 7-point response scale ranging from 0 (not at all confident) to 6 (completely confident). The score of PSEQ is the sum of all 10 items yielding score ranging from 0 to 60. The higher the score the stronger is self-efficacy belief.
Brief Pain Inventory | Pre-intervention, immediate post-intervention and 3 month post-intervention
  The Brief Pain inventory is a self-administrated questionnaire measures the severity and impact of the clinical pain. The questionnaire has four items for pain intensity and seven items for interference on general activity, mood, walking ability, normal walk, relations with other people sleep and enjoyment of life. The items for Pain are rated from 0 (no pain) to 10 (pain as bad as you imagine) and the items for interference are rated from 0 (does not interfere) to 10 (completely interfere). The pain score can be calculated by averaging the 4 items related to pain and the interference score can be calculated by averaging the 7 items related to interference. The higher the score, the more worsen of the condition.
Patient Specific Functional Scale | Pre-intervention, immediate post-intervention and 3 month post-intervention
  The Patient Specific Functional Scale is a self-reported questionnaire assessing the functional change of patients with musculoskeletal disorders. Subjects will ask to identify up to five important activities that have difficulty to perform and rate for the difficulty level of each identified activity on an 11-point scale ranging from "0" represents unable to perform to "10" represents able to perform. The Patient Specific Functional Scale score is the average score for the listed activities. The higher the score the more worsen of the condition.
Short Physical Performance Battery | Pre-intervention, immediate post-intervention and 3 month post-intervention
  The Short Physical Performance Battery is an objective measurement of the balance, lower extremity strength and functional capacity in elderly over 65 years of age. It includes three subscale of chair to stand tests, gait speed test and hierarchical balance test. Each test is scored from 0 (worst performance) to 4 (best performance). Adding together the three-subscale score yield the total score ranging from 0 to 12. The higher the total score the better the physical performance.
Patient satisfaction Survey | immediate post-intervention
  The patient satisfaction survey consists of 8 questions. One question concerns the compliance of exercise and rest of the seven questions concern the usefulness of the class. The subjects require rating from 0 (totally disagree) to 10 (totally agree) for their view to the questions. The questions include usefulness of the acceptance of pain concept, personalized goal setting, pamphlet, exercise taught, self-management concept, overall satisfaction, and overall improvement on back pain. The higher the score the higher the patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Man Ha Sharon Tsang, Doctor, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verhagen AP, Downie A, Popal N, Maher C, Koes BW. Red flags presented in current low back pain guidelines: a review. Eur Spine J. 2016 Sep;25(9):2788-802. doi: 10.1007/s00586-016-4684-0. Epub 2016 Jul 4. PMID 27376890
- [Background] National Guideline Centre (UK). Low Back Pain and Sciatica in Over 16s: Assessment and Management. London: National Institute for Health and Care Excellence (NICE); 2016 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK401577/ PMID 27929617
- [Background] Vadala G, Russo F, De Salvatore S, Cortina G, Albo E, Papalia R, Denaro V. Physical Activity for the Treatment of Chronic Low Back Pain in Elderly Patients: A Systematic Review. J Clin Med. 2020 Apr 5;9(4):1023. doi: 10.3390/jcm9041023. PMID 32260488
- [Background] Straube S, Harden M, Schroder H, Arendacka B, Fan X, Moore RA, Friede T. Back schools for the treatment of chronic low back pain: possibility of benefit but no convincing evidence after 47 years of research-systematic review and meta-analysis. Pain. 2016 Oct;157(10):2160-2172. doi: 10.1097/j.pain.0000000000000640. PMID 27257858
- [Background] Jacobs, C. (2015). Contextual pain management physiotherapy. NPUT center of St Thomas Hospital London UK.
- [Background] Godfrey E, Galea Holmes M, Wileman V, McCracken L, Norton S, Moss-Morris R, Pallet J, Sanders D, Barcellona M, Critchley D. Physiotherapy informed by Acceptance and Commitment Therapy (PACT): protocol for a randomised controlled trial of PACT versus usual physiotherapy care for adults with chronic low back pain. BMJ Open. 2016 Jun 7;6(6):e011548. doi: 10.1136/bmjopen-2016-011548. PMID 27267109
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Tsang, R. C. (2004). Measurement properties of the Hong Kong Chinese version of the Roland-Morris disability questionnaire. Hong Kong Physiotherapy Journal, 22(1), 40-49.
- [Background] McCracken LM. Committed action: an application of the psychological flexibility model to activity patterns in chronic pain. J Pain. 2013 Aug;14(8):828-35. doi: 10.1016/j.jpain.2013.02.009. Epub 2013 May 4. PMID 23651881
- [Background] Wong WS, McCracken L, Wong S, Chen PP, Chow YF, Fielding R. The Chinese version of the 8-item Committed Action Questionnaire (ChCAQ-8): A preliminary analysis of the factorial and criterion validity. Psychol Assess. 2016 Jun;28(6):e111-8. doi: 10.1037/pas0000187. Epub 2015 Jul 27. PMID 26214015
- [Background] Vowles KE, McCracken LM, McLeod C, Eccleston C. The Chronic Pain Acceptance Questionnaire: confirmatory factor analysis and identification of patient subgroups. Pain. 2008 Nov 30;140(2):284-291. doi: 10.1016/j.pain.2008.08.012. Epub 2008 Sep 27. PMID 18824301
- [Background] Liu Y, Wang L, Wei Y, Wang X, Xu T, Sun J. Validation of a Chinese version of the Chronic Pain Acceptance Questionnaire (CAPQ) and CPAQ-8 in chronic pain patients. Medicine (Baltimore). 2016 Aug;95(33):e4339. doi: 10.1097/MD.0000000000004339. PMID 27537558
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Lim HS, Chen PP, Wong TC, Gin T, Wong E, Chan IS, Chu J. Validation of the Chinese version of pain self-efficacy questionnaire. Anesth Analg. 2007 Apr;104(4):918-23. doi: 10.1213/01.ane.0000255731.24092.a5. PMID 17377107
- [Background] Poquet N, Lin C. The Brief Pain Inventory (BPI). J Physiother. 2016 Jan;62(1):52. doi: 10.1016/j.jphys.2015.07.001. Epub 2015 Aug 21. No abstract available. PMID 26303366
- [Background] Wang XS, Mendoza TR, Gao SZ, Cleeland CS. The Chinese version of the Brief Pain Inventory (BPI-C): its development and use in a study of cancer pain. Pain. 1996 Oct;67(2-3):407-16. doi: 10.1016/0304-3959(96)03147-8. PMID 8951936
- [Background] Stratford, P., Gill, C., Westaway, M., & Binkley, J. (1995). Assessing disability and change on individual patients: a report of a patient specific measure. Physiotherapy canada, 47(4), 258-263.
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Laerd Statisics. (2018). Mixed ANOVA using SPSS Statistics. Retrieved from https://statistics.laerd.com/spss-tutorials/mixed-anova-using-spss-statistics.php
- [Background] Lakens D. Calculating and reporting effect sizes to facilitate cumulative science: a practical primer for t-tests and ANOVAs. Front Psychol. 2013 Nov 26;4:863. doi: 10.3389/fpsyg.2013.00863. PMID 24324449